CLINICAL TRIAL: NCT05908331
Title: MagicTouch Sirolimus-coated Balloon for Treatment of In-Stent Restenosis in Coronary Artery Lesions
Brief Title: MagicTouch for Treatment of In-Stent Restenosis in Coronary Artery Lesions
Acronym: MAGICAL ISR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concept Medical Inc. (Industry)
Collaborators: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-US-R02
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: In-Stent Restenosis; Cardiovascular Diseases; Coronary Artery Disease
Keywords: Drug coated balloon; Sirolimus coated balloon; ISR; Magic Touch; SCB; Concept Medical; MAGICAL ISR
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: 2:1 randomized trial (MagicTouchTM vs. "plain old" balloon angioplasty [POBA])
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded till the primary endpoint of 12 months and the angiographic core laboratory will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- MagicTouch Sirolimus-Coated Balloon (Experimental): Magic TouchTM is a Sirolimus Coated Balloon catheter intended to be used in coronary applications, treats the atherosclerosis of the coronary arteries by eluting the immunosuppressant agent Sirolimus without leaving behind a metallic scaffold.
  Interventions: Device: Sirolimus Drug Coated Balloon
- POBA (Active Comparator): plain old balloon angioplasty
  Interventions: Device: Plan balloon Angioplasty (POBA)

INTERVENTIONS:
Device: Sirolimus Drug Coated Balloon — Magic TouchTM (Concept Medical) is a semi-compliant sirolimus drug coated balloon (SCB) for PCI, based on a polymer-free and nanocarrier based drug delivery technology.
  Arms: MagicTouch Sirolimus-Coated Balloon
Device: Plan balloon Angioplasty (POBA) — Plan balloon used to open clogged or narrow coronary arteries due to underlying atherosclerosis
  Arms: POBA

SUMMARY:
A Prospective, Multicenter, Randomized, Two-Arm, Single-blind Superiority Trial to Evaluate the Safety and Efficacy of the MagicTouch™ Sirolimus- Coated Balloon in the Treatment of Coronary Drug-Eluting Stent In-Stent Restenosis.

Subjects with prior DES implantation presenting with ISR lesions undergoing PCI will be randomized into two groups: treatment with the MagicTouch™ sirolimus-coated balloon or POBA on a 2:1 basis. Approximately 492 subjects will be enrolled in the randomized study in a maximum of 50 study sites located in the United States.

The goal is to establish the safety and efficacy of the MagicTouch™ sirolimus- coated balloon in treatment of coronary in-stent restenosis (ISR).

DETAILED DESCRIPTION:
All subjects providing informed consent will have their medical history reviewed and will undergo a physical examination, laboratory screen, and a standardized 12-lead ECG within 7 days of procedure. Women of childbearing potential will have a pregnancy test within one week prior to the procedure. If subjects meet the inclusion and exclusion criteria of the study, they will be randomized to one of two treatment groups, and will then undergo treatment with MagicTouch™ sirolimus-coated balloon or POBA of the target ISR lesion, per trial protocol.

One pre-procedure and all post-procedure biomarker blood draws will be sent to a central core laboratory for analysis of troponin T. Evaluation of post-procedural biomarker blood draws in local laboratories are not mandated but may be performed as part of standard of care.

During the index hospitalization, patients will undergo a clinical assessment and 12-lead ECG; and they will have cardiac biomarkers drawn before the intervention to establish baseline biomarker level and confirmation that the biomarkers are falling. At least one post procedure biomarker (core lab) will be drawn at a minimum of 4 hours after PCI as part of the assessment of periprocedural myocardial infarction and significant periprocedural myocardial injury (at 6-8 hour intervals depending on whether the patient remains admitted). If no procedural complications have occurred and there are no signs of ischemia on post-procedure ECG or clinical assessment, the patient may be discharged per local practice and no additional biomarker levels need to be drawn (beyond the protocol-mandated core laboratory draw at a minimum of 4 hours). If the patient remains admitted cardiac biomarkers (core lab) should be drawn every 6-8 hours until at least 2 total post-procedural core laboratory biomarker draws have passed or clinical standard-based biomarker levels have peaked per local labs or the patient is discharged.

After hospital discharge, subjects will be followed at 30 days (+1 week), 6 months (+2 weeks), and 12 months (+1 month) and then 24, 36, 48 and 60 months (+1 month) post procedure. Yearly vital status information will be collected by telephone follow-up. At the 12-month visit, subjects will undergo 12-lead ECG, blood count, coagulation profile and blood chemistry tests. New and ongoing AEs and concomitant medications will also be assessed.

All elective angiograms performed on the target vessel during the 12-month follow-up period should be preceded by a physician evaluation, during which the physician will indicate whether the subject's clinical status warrants revascularization, i.e. the subject has clinical evidence of ischemia. All films, including unscheduled angiograms, are to be sent to the angiographic core laboratory for review. The angiographic core laboratory will be blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject (or legal guardian) understands the trial requirements and treatment procedures and provides written informed consent prior to any trial-specific tests or treatment
3. Patient with an indication for PCI due to suspected in-stent restenosis
4. Non-target lesion PCI are allowed in non-target vessels to be treated with approved interventional devices prior to randomization as follows:

Angiographic Inclusion Criteria:

1. In-stent restenosis after drug-eluting stent implantation(s) in the target lesion (i.e. single and multiple stent layer ISR cases are eligible)
2. Target lesion must have visually estimated stenosis ≥50% and less than 100% diameter stenosis in symptomatic patients; or a visually estimated target lesion diameter stenosis of ≥70%, or by evidence of ischemia by coronary physiology (fractional flow reserve [FFR] ≤0.80 or non-hyperemic pressure ratio [NHPR] ≤0.89) in absence of symptoms
3. Successful lesion preparation (residual stenosis <30%), without complications (no or slow flow, flow-limiting dissection, perforation, distal embolization) and without plan for stenting
4. Target lesion in a native coronary artery
5. Thrombolysis In Myocardial Infartction (TIMI) grade flow ≥1 in target lesion
6. Target reference vessel diameter (visual estimation) >2.0 and ≤4.0 mm
7. Target lesion length (including tandem lesions) ≤36.0 mm (visual estimation) and can be covered by only one balloon
8. One ISR target lesion (overlapping stents are allowed) to be treated per patient and in single major coronary artery or side branch (reference vessel diameter >2.0 mm)
9. Other coronary lesions (ISR or non-ISR) in non-target vessel are allowed and may be treated by any approved interventional device, but must be treated successfully prior to randomization

Exclusion Criteria:

General Exclusion Criteria (all must be absent for the patient to be eligible):

1. STEMI within 72 hours of presentation to the first treating hospital, whether a transfer facility or the study hospital
2. NSTEACS in whom the biomarkers have not peaked
3. PCI within the 24 hours prior to the index procedure (not including PCI performed in non-target lesions during the index procedure)
4. Prior DCB treatment (coronary or off-label peripheral) of target lesion ISR
5. Cardiogenic shock (defined as persistent hypotension [systolic blood pressure <90 mm Hg] or requiring vasoactive or hemodynamic support, including IABP)
6. Subject is intubated
7. Known left ventricular ejection fraction <30%
8. Relative or absolute contraindication to DAPT for at least 1 month (e.g., planned surgeries that cannot be delayed)
9. Subject has an indication for chronic oral anticoagulation treatment and a contraindication for concomitant treatment with a P2Y12 inhibitor
10. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6F sheath
11. Hemoglobin <9 g/dL
12. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3
13. White blood cell count <3,000 cells/mm3
14. Active infection undergoing treatment
15. Clinically significant liver disease
16. Renal insufficiency as defined by estimated glomerular filtration rate (eGFR) to be <30ml/min by the MDRD formula
17. Active peptic ulcer or active bleeding from any site
18. Bleeding from any site requiring active medical attention within the prior 8 weeks
19. History of bleeding diathesis or coagulopathy or likely to refuse blood transfusions
20. Cerebrovascular accident (CVA) within 3 months or has any permanent neurological defect as a result of CVA
21. Known allergy to the study device components or protocol-required concomitant medications:

    - sirolimus (as well as other limus drugs, analogues, or similar compounds), aspirin, clopidogrel and prasugrel and ticagrelor, heparin and bivalirudin, or iodinated contrast that cannot be adequately pre-medicated
22. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduce life expectancy to <24 months (e.g. cancer, heart failure, lung disease, severe valvular disease)
23. Patient is participating in or plans to participate in any other investigational drug or device trial that has not reached its primary endpoint
24. Women who are pregnant or breastfeeding (women of child-bearing potential must have a negative pregnancy test within one week before index procedure)
25. Women who intend to become pregnant within 12 months after the index procedure
26. Patient has received an organ transplant or is on a waiting list for an organ transplant
27. Patient has received chemotherapy within 30 days before the index procedure or scheduled to receive chemotherapy any time after the index procedure
28. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease. Inhaled steroid and steroid use for contrast- allergy prophylaxis or treatment are allowed

Angiographic Exclusion Criteria (visual estimate) (all must be absent for the patient to be eligible):

1. More than 1 ISR lesion in the target vessel in segments that cannot be treated by a single 40mm length DCB (see Angiographic Inclusions #5 and #6 above)
2. ISR lesion in the target vessel in a segment that corresponds to a previously established/documented bare metal stent (BMS)
3. Unprotected left main lesions >50% or left main intervention
4. Primary PCI for STEMI
5. Coronary artery disease judged more suitable for surgical revascularization per guidelines and local heart team discussion
6. Another lesion in either the target vessel or non-target vessel is present that requires or has a high probability of requiring PCI within 12 months after the index procedure
7. Prior brachytherapy or DCB treatment of target lesion
8. Target lesion is a bifurcation restenosis involving both branches of a bifurcation in which the side branch reference vessel diameter is >2.0 mm
9. Target lesions located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
10. Target lesion contains large thrombus
11. Target lesion is heavily calcified
12. Target lesion is a chronic total occlusion (or subtotal) without adequate lesion preparation.* Total and subtotal occlusions may be enrolled assuming they can be crossed with a wire and demonstrate TIMI grade 3 flow at the time of randomization.
13. Diffuse distal disease to target lesion with impaired runoff

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
TLF (Target Lesion Failure) | 12 months
  The composite rate of cardiac death, target-vessel MI (Myocardial Infarction) or ischemia-driven TLR (Target Lesion Revascularization)

SECONDARY OUTCOMES:
MACE (Major adverse cardiovascular events) | 30 days and 6, 12, 24, 36, 48, and 60 months
  composite of cardiovascular mortality, any MI (Myocardial Infarction), and ID-TLR (Ischemia-Driven Target Lesion Revascularization)
TVF (Target vessel failure) | 30 days and 6, 12, 24, 36, 48, and 60 months
  composite of cardiovascular mortality, ID-TVR (Ischemia-Driven Target Vessel Revascularization), and TV-MI (Target Vessel Myocardial Infarction)
Any revascularization | 30 days and 6, 12, 24, 36, 48, and 60 months
  any repeat PCI or CABG
ID-TLR (Ischemia-Driven Target Lesion Revascularization) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Repeat revascularization of the target lesion due to recurrent ischemia
TLR (Target Lesion Revascularization) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Repeat revascularization of the target lesion
ID-TVR (Ischemia-Driven Target Vessel Revascularization) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Repeat revascularization of the target vessel due to recurrent ischemia
TVR (Target Vessel Revascularization) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Repeat revascularization of the target vessel
All-cause mortality | 30 days and 6, 12, 24, 36, 48, and 60 months
  Death from any cause
Cardiovascular mortality | 30 days and 6, 12, 24, 36, 48, and 60 months
  Death due to coronary artery disease or complications of coronary treatment
Any MI (Myocardial Infarction) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Any Myocardial Infarction
TV-MI (Target Vessel Myocardial Infarction) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Myocardial Infarction related to the target vessel
Q-wave MI (Myocardial Infarction) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Myocardial Infarction demonstrated by new pathological Q waves on ECG
Non-Q-wave MI (Myocardial Infarction) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Myocardial Infarction not demonstrated by new pathological Q waves on ECG
Cardiovascular mortality or MI (Myocardial Infarction) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Either cardiovascular death or any Myocardial Infarction
All-cause mortality or MI (Myocardial Infarction) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Either death from any cause or any Myocardial Infarction
All-cause mortality, MI (Myocardial Infarction), or TVR (Target Vessel Revascularization) | 30 days and 6, 12, 24, 36, 48, and 60 months
  Death from any cause, any Myocardial Infarction, or Target Vessel Revascularization
Any definite or probable target lesion stent thrombosis by ARC (Academic Research Consortium) criteria | 30 days and 6, 12, 24, 36, 48, and 60 months
  Definite or probable stent thrombosis in the target lesion according to the ARC (Academic Research Consortium) definition
Probable target lesion stent thrombosis by ARC (Academic Research Consortium) criteria | 30 days and 6, 12, 24, 36, 48, and 60 months
  Probable stent thrombosis in the target lesion according to the ARC definition
Definite target lesion stent thrombosis by ARC (Academic Research Consortium) criteria | 30 days and 6, 12, 24, 36, 48, and 60 months
  Definite stent thrombosis in the target lesion according to the ARC definition
BARC (Bleeding Academic Research Consortium) type 3-5 bleeding | 30 days and 6, 12, 24, 36, 48, and 60 months
  Significant or severe bleeding according to the BARC definition
Procedure Success | 30 days and 6, 12, 24, 36, 48, and 60 months
  ability to deliver the device and achieve a less than 30% residual stenosis by QCA (quantitative coronary angiography) without major complication or bailout stenting

OTHER OUTCOMES:
Angina as assessed by SAQ-7 (Seattle Angina Questionnaire) | 30 days, 6, 12, 24, 36, 48 and 60 months
  Quality of Life Endpoint, Angina will be assessed at these specified timepoints and prior to any invasive procedure

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Cardiology, PC - Princeton Baptist Medical Center, Birmingham, Alabama
  - Dignity Health - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Cedars - Sinai Medical Center, Los Angeles, California
  - Yale University / Yale New Haven Hospital, New Haven, Connecticut
  - Cheek-Powell Heart and Vascular Pavilion, Clearwater, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - The Cardiac & Vascular Institute Research Foundation, Gainesville, Florida
  - Tampa General Hospital / University of South Florida, Tampa, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Metropolitan Heart and Vascular Institute, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - VA New York Harbor Healthcare System, New York, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma University Health (OU Health), Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Prisma Health, Greenville, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Baylor Scott and White Heart and Vascular Hospital, Dallas, Texas
  - Baylor Scott & White - The Heart Hospital - Plano, Plano, Texas
  - West Virginia University and Vascular Institute, Morgantown, West Virginia